CLINICAL TRIAL: NCT05295316
Title: Risk Factors Recognition of Primary Fibromyalgia: a Case-control Study
Brief Title: Risk Factors of Primary Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Studio Osteopatico Busto Arsizio (Other)
Responsible Party: Principal Investigator, Carolina Lavazza, Osteopath, Studio Osteopatico Busto Arsizio
Other Study IDs: 230176
Record Dates: First submitted 2022-03-11; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Fibromyalgia
Keywords: Osteopathy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia: FM group was recruited at AMaR (rheumatic patients association of Piedmont) and the diagnosis of primary fibromyalgia was confirmed by the referring rheumatologist of the AMaR association.
  Interventions: Other: Life Stressor Checklist Revised (LSC-R) (Appendix 1)
- Control: The control group was recruited in the same geographic area as the FM participant. The general practitioner of each individual patient certified the subject's state of good health.
  Interventions: Other: Life Stressor Checklist Revised (LSC-R) (Appendix 1)

INTERVENTIONS:
Other: Life Stressor Checklist Revised (LSC-R) (Appendix 1) — Evaluation of stress factor as risk factor for fibromyalgia development

SUMMARY:
Fibromyalgia (FM) is a condition with a different non-specific symptoms which lead to a difficult diagnosis. Study suggests that osteopathy can help in improving FM symptoms, nevertheless, it can be difficult to identify which patients may benefit. The knowledge of FM risk factor can be useful tool for osteopaths and other clinician to implement a targeted, fast and multidisciplinary treatment protocol for those kind of patient.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* Patient from Piedmont
* age between 20 and 65 years old
* inform consent
* for case group primary or secondary fibromyalgia

Exclusion Criteria:

* systemic or rheumatic or neoplastic diseases
* for control group the presence of primary or secondary fibromyalgia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female women were used because have higher risk of fibromyalgia development.
Study Population: Female patients with or without fibromyalgia
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Incidence of 29 stressing events | 1 year
  The LSC-R questionnaire was used to evaluate the incidence of each stressor event

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Lavazza, MSc, Study Chair — Accademia Italiana Medicina Osteopatica
Locations (1):
- OsteoMedical, Novara, Italy

IPD SHARING:
Plan to Share IPD: No